CLINICAL TRIAL: NCT07216378
Title: On Demand Treatment of Angioedema Attacks in Pediatric (Ages 2-11) Post-Trial and Naive Patients With Hereditary Angioedema (HAE) With Sebetralstat
Brief Title: Treatment of Angioedema Attacks in Pediatric (Ages 2-11) Post-Trial and Naive Patients With HAE With Sebetralstat
Status: Available | Type: Expanded Access
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KVD900-EAP-US-2
Record Dates: First submitted 2025-09-12; First posted 2025-10-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — sebetralstat

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Sebetralstat — Oral Plasma Kallikrein Inhibator
  Other Names: KVD900

SUMMARY:
The sebetralstat Early Access Program (EAP) provides early access to the investigational medicinal product (IMP) sebetralstat to eligible and approved Hereditary Angioedema (HAE) pediatric (ages 2-11) post-trial and naïve patients for the on-demand treatment of angioedema attacks where the treating Physician determines they might benefit from this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 2 to 11 years of age.
* Parent or LAR provides signed informed consent and patient provides assent (when applicable).
* Confirmed diagnosis of HAE.

Exclusion Criteria:

* Confirmed diagnosis of HAE with nC1-INH or acquired angioedema
* Patient weighs <9.5 kg
* Patient participated in the KVD900-303 trial and withdrew prior to trial completion per the protocol or trial closure
* Any clinically significant medical condition or medical history that, in the opinion of the Treating Physician, would interfere with the patient's safety.
* Known hypersensitivity to sebetralstat or its excipients.
* Patient with a medical history or known to have severe hepatic impairment (Child Pugh C).
* Patients who require sustained use of strong cytochrome P450 3A4 inhibitors or inducers.

Ages: 2 Years to 11 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - KalVista Investigative Site, Evansville, Indiana
  - KalVista Investigative Site, Wheaton, Maryland
  - KalVista Investigative Site, St Louis, Missouri